CLINICAL TRIAL: NCT05666765
Title: Comparative Study Between the Effect of Isotretinoin, Silymarin and Their Combination in the Treatment of Patients With Acne Vulgaris
Brief Title: Comparison Between Isotretinoin, Silymarin and Both in the Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ghada mohamed abdelmonem mohamed Tantawy, Principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treatment of acne vulgaris
Record Dates: First submitted 2022-12-08; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Prospective controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- acne vulgaris patients group 1 (Experimental): acne patients will be rondomly assigned to 1 of the 3 interventions (isotretinoin, silymarin, or both)
  Interventions: Drug: Isotretinoin ,silymarin
- acne vulgaris patients group 2 (Experimental): acne patients will be rondomly assigned to 1 of the 3 interventions (isotretinoin, silymarin, or both)
  Interventions: Drug: Isotretinoin ,silymarin
- acne vulgaris patients group 3 (Experimental): acne patients will be rondomly assigned to 1 of the 3 interventions (isotretinoin, silymarin, or both)
  Interventions: Drug: Isotretinoin ,silymarin

INTERVENTIONS:
Drug: Isotretinoin ,silymarin — 20mg/day isotretinoin for 3 months. 140 mg/day silymarin for 3 months. 20mg/day isotretinoin and 140mg/day silymarin for 3 months.

SUMMARY:
This study aims to compare the effects of isotretinoin and silymarin or both in treatment of acne and their effects on the level of IGF-1, SAA1 and malondialdehyde (MDA) in acne patients.

DETAILED DESCRIPTION:
Acne vulgaris, a common and chronic disorder of the pilosebaceous unit, affects up to 85% of adolescent and young adults. The pathogenesis of acne is multifactorial. Traditionally, four distinct processes were believed to play critical roles: increased sebum production, alteration of keratinization processes leading to comedone formation, follicular colonization by Propionibacterium acnes (P.acnes) and inflammatory mediators around pilosebaceous unit.

Orally administered isotretinoin is currently the only agent that can affect all four main factors implicated in acne.

Serum insulin-like growth factor -1(IGF)-1 is a polypeptide hormone that has effects on sebocyte differentiation and proliferation. It leads to lipogenesis, and synthesis of inflammatory cytokines. IGF-1 also stimulates androgen synthesis leading to overproduction of sebum.

Propionibacterium acnes can increase the release of serum amyloid A1 (SAA1) .There is significant elevation of SAA1 in patients with acne, with a positive correlation with its severity.

Oxidative stress plays a role in the pathogenesis of acne in part due to the generation of reactive oxygen species (ROS) in response to infection by the bacterium Propionibacterium acnes, which colonizes the skin and grows in plugged hair follicles, thus attracting inflammatory cells, mainly neutrophils. These in turn secrete inflammatory mediators and generate ROS, which augments the inflammatory response and tissue damage.

Silymarin, the main active component of milk thistle consists of a mixture of flavonolignans and flavonoid taxifolin. Silymarin acts as a hepatoprotective, anticancer, anti-inflammatory and immunomodulatory agent.

Silymarin acts as a free radical scavenger, stabilizes the plasma membrane and reduces the production of inflammatory mediators produced by P. acnes, and scavenges the released free radicals.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years or more. Patient with moderate or severe acne. Not receiving acne treatment in the last month.

Exclusion Criteria:

* Pregnancy or lactation. Patients with known hypersensitivity to isotretinoin or silymarin. Patients with depression, liver diseases or high cholesterol. Patients with acromegaly. Patients with chronic inflammatory, infective or neoplastic disorders.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Global Acne Grading Classification | 3 months
  Global Acne Grading System (GAGS) Each is derived by multiplying the factors-2 for forehead, 2 for each check, 1 for nose, 1 for chin, 3 for both chest and back by the most heavily weighted lesion within each region (1 for ≥ one comedone, 2 for ≥ one papule,3 for ≥ one pustule, and 4 for ≥ one nodule).

SECONDARY OUTCOMES:
Liver function tests | 3 months
  Serum AST and ALT measure before and after 3 months therapy
Lipid profile | 3 months
  serum cholesterol, TG, LDL and HDL levels in blood before and after 3 months therapy
Insulin growth factor -1 | 3 months
  Assessment of IGF-1 level in blood before and after 3 months therapy
serum amyloid A1 | 3 months
  Assessment of serum amyloid A1 level before and after 3 months therapy
Malondialdehyde | 3 months
  Assessment of Malondialdehyde level in blood before and after 3 months therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ghada F Hassan, A.professor, Study Chair — Tanta University; Dalia R Elafify, Doctor, Study Chair — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hazarika N. Acne vulgaris: new evidence in pathogenesis and future modalities of treatment. J Dermatolog Treat. 2021 May;32(3):277-285. doi: 10.1080/09546634.2019.1654075. Epub 2019 Aug 29. PMID 31393195
- [Background] Shie Morteza M, Hayati Z, Namazi N, Abdollahimajd F. Efficacy and safety of oral silymarin in comparison with oral doxycycline and their combination therapy in the treatment of acne vulgaris. Dermatol Ther. 2019 Nov;32(6):e13095. doi: 10.1111/dth.13095. Epub 2019 Oct 21. PMID 31579978